CLINICAL TRIAL: NCT02073825
Title: Web Intervention for Concerned Partners to Prevent Service Member Alcohol Abuse
Brief Title: Web Intervention for Concerned Partners to Prevent Service Member Alcohol Abuse Abuse
Acronym: PC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RAND (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Karen Osilla, Behavioral Scientist, RAND
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R34AA023123 (NIH); R34AA023123 (NIH)
Record Dates: First submitted 2014-02-20; First posted 2014-02-27 (Estimated); Last update posted 2017-09-29 (Actual); Status verified 2017-09

CONDITIONS: Alcohol Abuse
Keywords: Computer-assisted interventions; Alcohol use disorders; At-risk drinking; Spouses; Military; Brief Intervention
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Web Brief Intervention (WBI) (Experimental): 4-session WBI
  Interventions: Behavioral: Web Brief Intervention (WBI)
- Delayed-WBI (No Intervention): 4-session WBI after follow-up

INTERVENTIONS:
Behavioral: Web Brief Intervention (WBI) — 4-session WBI
  Arms: Web Brief Intervention (WBI)

SUMMARY:
The purpose of this study is to adapt and pilot-test a web-based intervention intended to help concerned partners provide support to service members with alcohol misuse and to begin development of a service member module based on service member's input.

DETAILED DESCRIPTION:
U.S. military service members engaged in alcohol misuse are a vulnerable population with high unmet need. Alcohol misuse is a stage of problem drinking that occurs before abuse and dependence, placing service members' partners and families at risk for serious consequences. Unfortunately, existing military reporting policies may discourage service members from seeking help for fear of negative career consequences. Service members report encouragement from their partners as the most prevalent facilitator of seeking care and individuals who change their drinking patterns most often cite partner support as the most helpful mechanism in supporting change. Thus, targeting service members' partners using preventive interventions can be an important vehicle for preventing the progression to abuse and dependence. A 3-year study is proposed to adapt and pilot-test a web-based intervention (WBI) intended to help concerned partners (CPs) provide support to service members with alcohol misuse and to begin development of a service member module based on service member's input. First, an evidence-based intervention known as Community Reinforcement and Family Training (CRAFT) intervention will be adapted to the web. The specific aims are as follows: Aim 1: Develop a 4-session web-based intervention (WBI) prototype and make iterative revisions based on feedback from 15-20 CPs. Aim 2: Conduct a randomized controlled pilot-test of the finalized WBI (n=50) compared to delayed WBI (n=50), and evaluate the impact of the WBI on CP's reports of service member help-seeking (e.g., counseling, self-help, primary care, treatment) and drinking, and CP well-being and relationship satisfaction three months after the intervention. Aim 3: Begin development of a follow-on WBI module for service members based on service member input and content evaluation. Service members will be asked their intervention preferences and feedback on a proposed WBI for them. This project is significant because it has the potential to benefit a large population of military service members who may be disproportionately affected by the current OEF/OIF/OND conflicts and whose drinking misuse would otherwise go undetected and untreated. It also develops a new prevention model that does not rely on service members or partners attending a hospital or clinical facility to access care. The proposed study is innovative because there are no CP-based preventive interventions addressing misuse. This pilot study will inform the development of an R01 trial that evaluates a larger randomized study of a WBI for CPs with a follow-on intervention for service members.

ELIGIBILITY:
Inclusion Criteria:

1. if they are currently living with their partner,
2. if they have had contact with their partner at least 40% of the time in the past 90 days (e.g., most of the evenings or most of the days in a given week),
3. if they are in a romantic relationship with the service member,
4. if they have a computer they can use in a private area,
5. if the CP and service member are at least 18 years of age,
6. if their partner is currently an active duty service member,
7. if the CP or service member has not attended couples or drug/alcohol counseling in the past 60 days,
8. if the CP does not plan to separate from their partner in the next 60 days,
9. if they feel their partner has a problem with their drinking, and
10. if they do not endorse any domestic violence in the past year. -

Exclusion Criteria:

1. if the CP plans to seek counseling in the next 90 days, and/or
2. reports feeling unsafe to discuss drinking with his/her partner -

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 312 (Actual)
Dates: Start 2014-11; Primary Completion 2015-10 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
Perceptions of Partner's Drinking | Three months after intervention
  DNRF: "Consider a typical week during the past month (30 days). How much alcohol, on average, (measured in number of drinks), do you think your partner had on each day of a typical week?"
Concern about Partner's Drinking | Three months after intervention
  Thinking about your Partner's Drinking (TPD): http://www.sciencedirect.com/science/article/pii/S0306460313002517
Partner's readiness to change | Three months after intervention
  On a scale from 0 to 10, how ready do you feel your partner is to change his/her drinking?
Partner help-seeking | Three months after intervention
  On a scale from 0 to 10, how ready do you think your partner feels about seeking help for their drinking (for example, talking with a counselor or going to AA meetings regularly).
Relationship Quality | Three months after intervention
  Quality Marriage Index (QMI): Norton, R. (1983). Measuring marital quality: A critical look at the dependent variable. Journal of Marriage and Family, 45, 141-151.

SECONDARY OUTCOMES:
CP Depression and Anxiety | Three months after intervention
  PHQ-8 and BAI
Family Environment | Three months after intervention
  Family Environment Scale (FES)

CONTACTS AND LOCATIONS:
Overall Officials: Karen C Osilla, PhD, Principal Investigator — RAND
Locations (1):
- RAND, Santa Monica, California, United States

REFERENCES:
- [Background] Osilla KC, Pedersen ER, Gore K, Trail T, Howard SS. Study design to develop and pilot-test a web intervention for partners of military service members with alcohol misuse. Addict Sci Clin Pract. 2014 Sep 2;9(1):18. doi: 10.1186/1940-0640-9-18. PMID 25179672
- [Background] Osilla KC, Pedersen ER, Tolpadi A, Howard SS, Phillips JL, Gore KL. The Feasibility of a Web Intervention for Military and Veteran Spouses Concerned About Their Partner's Alcohol Misuse. J Behav Health Serv Res. 2018 Jan;45(1):57-73. doi: 10.1007/s11414-016-9546-3. PMID 28039559
- [Background] Pedersen, E. R., Osilla, K. C., Helmuth, E. D., Tolpadi, A., & Gore, K. (2017). Reaching Concerned Partners of Heavy Drinking Service Members and Veterans through Facebook. Military Behavioral Health, 5:3, 265-273, DOI: 10.1080/21635781.2017.1316804
- [Result] Rodriguez LM, Osilla KC, Trail TE, Gore KL, Pedersen ER. Alcohol Use Among Concerned Partners of Heavy Drinking Service Members and Veterans. J Marital Fam Ther. 2018 Apr;44(2):277-291. doi: 10.1111/jmft.12261. Epub 2017 Aug 7. PMID 28782116
- [Derived] Trail TE, Osilla KC, Rodriguez LM, Pedersen ER, Gore KL. Exploring the association between changes in partner behaviors, perceived service member drinking, and relationship quality: Secondary analysis of a web-based intervention for military partners. J Subst Abuse Treat. 2019 Mar;98:66-72. doi: 10.1016/j.jsat.2019.01.002. Epub 2019 Jan 3. PMID 30665606